CLINICAL TRIAL: NCT03068000
Title: Effect of Judo Training Compared to Ball Games on Motor Skills, Physical Fitness, Quality of Life and Cardiovascular Parameters in Children and Adolescents: Randomized Crinical Trial
Brief Title: Effect of Judo Training Compared to Ball Games on Motor Skills, Physical Fitness, Quality of Life and Cardiovascular Parameters in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Bruna Thamyres Ciccotti Saraiva, Master's Degree Student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 26702414.0.0000.5402
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Child Behavior; Adolescent Behavior
Keywords: Martial arts; Judo; Motor skills; Physical fitness; Cardiovascular parameters; Quality of life; Physical Activity
MeSH Terms: conditions — Child Behavior; Adolescent Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Judo training and Ball games
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the evaluators will be blind as well as the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Judo training (Experimental): Judo intervention will take place twice a week, lasting 50 minutes per session, for 3 months, divided into general exercises: warm-up and stretching specific to the sport; Specific exercises of the sport: shock absorption, falls cushioning (Ukemi-waza), immobilization techniques (hon-kesa-gatame and tate-shiho-gatame) and projection (o-soto-gari, o-goshi, ashi-guruma, koshi-guruma, tai-otoshi and others); And fight simulation: randori.
  Interventions: Behavioral: Judo Training
- Ball games (Active Comparator): The Ball Games will take place twice a week, with a duration of 50 minutes per session, for 3 months, divided into general exercises: heating and specific stretching with ball; Specific exercises of the sport: fundamentals of sports with ball, exercises with ball; And games: games will be given at the end of the lesson to work out all the fundamentals and specific exercises in general.
  Interventions: Behavioral: Ball Games

INTERVENTIONS:
Behavioral: Judo Training — Judo intervention is divided into general exercises: warm-up and stretching specific to the sport; Specific exercises of the sport: shock absorption, falls cushioning (Ukemi-waza), immobilization techniques (hon-kesa-gatame and tate-shiho-gatame) and projection (o-soto-gari, o-goshi, ashi-guruma, koshi-guruma, tai-otoshi and others); And fight simulation: randori.
  Arms: Judo training
Behavioral: Ball Games — The Ball Games is divided into general exercises: heating and specific stretching with ball; Specific exercises of the sport: fundamentals of sports with ball, exercises with ball; And games: games will be given at the end of the lesson to work out all the fundamentals and specific exercises in general.
  Arms: Ball games

SUMMARY:
There will be a three-month intervention with two groups: judo training and ball games, twice a week, for 50 minutes. The sample will consist of children and adolescents with low socioeconomic status, participants of a philanthropic institution, aged between 6 and 15 years, who will be randomized in the two groups mentioned above. Motor skills, physical fitness, cardiovascular parameters and questionnaire assessing socioeconomic status, quality of life, physical activity level, screen time, sleep quality, back pain, food intake and body image dissatisfaction will be evaluated.

DETAILED DESCRIPTION:
The sample will be of 66 participants, randomized into two groups 33 in judo and 33 in ball games. According to the sample calculation based on the study of Bala and Drid (2010) title "Anthropometric and Motor Features of Young Judoists in Vojvodina", who analyzed motor skills in young judokas and untrained control, using the variable slalom with 3 balls (functional coordination and the age group from 11 to 13 years. In which the difference between the means was of 36.86 and the standard deviation of 53.78, with the power of the 80% test and significance of 5% in boys. In girls the sample calculation was the same number (33 for group) using the same variable slalom with 3 balls (functional coordination and the some age group from 11 to 13 years, the difference between the means was 10.45 and the standard deviation of 15.05, with the power of the 80% test and significance of 5%

The present study was approved by the Research Ethics Committee of FCT/UNESP (CAAE: 26702414.0.0000.5402), with the number of opinion 549.549.

Interventions

Judo Training Judo intervention will take place twice a week, lasting 50 minutes per session, divided into general exercises: warm-up and stretching specific to the sport; Specific exercises of the sport: shock absorption, falls cushioning (Ukemi-waza), immobilization techniques (hon-kesa-gatame and tate-shiho-gatame) and projection (o-soto-gari, o-goshi, ashi-guruma, koshi-guruma, tai-otoshi and others); And fight simulation: randori.

Ball Games The Ball Games will take place twice a week, with a duration of 50 minutes per session, divided into general exercises: heating and specific stretching with ball; Specific exercises of the sport: fundamentals of sports with ball, exercises with ball; And games: games will be given at the end of the lesson to work out all the fundamentals and specific exercises in general.

Statistical Analysis We will perform the Shapiro-Wilks normality test, analysis of variance (ANOVA) of repeated measures and the effect size will be calculated by Eta Squared, all using SPSS Software version 13.0 and adopting a significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled in the philanthropic institution;
* Be between 6 and 15 years old;
* Study at the opposite time to the project, in which the intervention will occur;
* To present a free and informed consent form signed by parents and/or guardians.

Exclusion Criteria:

* Do not take any type of medication that influences the evaluated variables;
* Do not present any type of orthopedic problem that prevents the accomplishment of the activities;
* Not being pregnant.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Equilibrium | Baseline and three months of follow up
  The motor skills will be by means of the Körperkoordination Test für Kinder (KTK) (Kiphard, Schilling, 1974) test battery consisting of four stations, and Equilibrium Beam is one, in which the evaluated one must walk on backs of three different widths, measured in how many steps on the toolbar.

SECONDARY OUTCOMES:
Change of Quality of Life | Baseline and three months of follow up
  Quality of life was assessed by the KIDSCREEN-52 questionnaire validated by Guedes and Guedes (2011) for children and adolescents offering information on health-related quality of life.
Change of Lateral Jumping | Baseline and three months of follow up
  The motor skills will be by means of the Körperkoordination Test für Kinder (KTK) (Kiphard, Schilling, 1974) test battery consisting of four stations: Lateral Jumping is one, consisting of the execution of the maximum of lateral jumps in 15 seconds, measured in number of jumps.
Change of Platform Transfer | Baseline and three months of follow up
  The motor skills will be by means of the Körperkoordination Test für Kinder (KTK) (Kiphard, Schilling, 1974) test battery consisting of four stations: Platform Transfer the maximum transfers in 20 seconds.
Change of Monopedal jump | Baseline and three months of follow up
  The motor skills will be by means of the Körperkoordination Test für Kinder (KTK) (Kiphard, Schilling, 1974) test battery consisting of four stations: Monopedal jump is one, in which the child jumps with one leg at a time trying to reach the maximum height, measured by means of a score adding the score of the two legs.
Change of Heart Rate | Baseline and three months of follow up
  Heart rate will be measured using an Omron oscillometric device validated for this population (Zanuto et al., 2016), measured in beats per minute (bpm).
Change of Blood Pressure | Baseline and three months of follow up
  Systolic and diastolic blood pressure will be measured using an Omron oscillometric device validated for this population (Christofaro et al., 2009), measured in millimeters of mercury (mmHg).
Change of Heart Rate Variability | Baseline and three months of follow up
  he heart rate variability was evaluated by means of a Polar frequency meter model RS800, in which it measures linear time and frequency domains and nonlinear domains such as the Poincaré Plot.
Change of Agility | Baseline and three months of follow up
  Agility will be measured by means of the Shuttle Run test, measured in seconds.
Change of Strenght of upper limbs | Baseline and three months of follow up
  The strength of upper limbs by force on the bar, measured in repetitions.
Change of Manual gripping force | Baseline and three months of follow up
  The manual gripping force by means of the dynamometer, measured in Kilograms.
Change of Abdominal strenght | Baseline and three months of follow up
  Agility will be measured by means of the Shuttle Run test, the strength of upper limbs by force on the bar, as well as the manual gripping force by means of the dynamometer, The abdominal strength with the one minute test the maximum number of repetitions.
Change of Strenght of legs | Baseline and three months of follow up
  The vertical and horizontal jumping is used to assess the strength of legs, measured in centimeters.
Change of Screen Time | Baseline and three months of follow up
  The screen time will be measured by six questions about how many hours the individual spends playing video games, using cell phones, computer or internet and television sitting during the week and the weekend.
Change of Back Pain | Baseline and three months of follow up
  Back pain will be evaluated using questionnaire, which asks if there is pain, tingling or numbness in the last year both in the upper and lower back and if it is impossible to perform the activities A health professional because of the pain and felt that pain in the last week. As well as for a pain scale of 0 to 10, if the individual presents pain.
Change of Sleep Quality | Baseline and three months of follow up
  The time of sleep, hours of sleep and quality of sleep will be evaluated by means of the mini sleep questionaire, in which it sees the frequency in which the individual presents problems in sleep, by score, being the lowest quality And higher lower quality sleep.
Change of Body Image Dissatisfaction | Baseline and three months of follow up
  Body image dissatisfaction will be assessed through the silhouettes scale for children and adolescents proposed by Kakeshita et al. (2009), in which it presents 11 figures from the smallest to the largest silhouette. With questions like: "Which picture represents your current body?" "Which of these figures represents the body you would like to have?" And "Which figure represents the ideal body for your gender?"
Socioeconomic Condition | Baseline and three months of follow up
  The questionnaire of the Brazilian Association of Research Companies (ABEP) to analyze the socioeconomic level and the educational level of the parents will be applied in adolescents.
Change of Food Intake | Baseline and three months of follow up
  Will be questioned how many days of the week in numbers the individual consumes fruits, vegetables and vegetables, dairy, fried, sweets, grains, white meat, soft drinks and snacks.
Physical Activity Level | Baseline and three months of follow up
  The questionnaire of Baecke et al. (1982) will analyze individual habits by measuring the level of physical activity in different domains

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Validation of Kakeshita scale — http://scielo.br/pdf/ptp/v25n2/a15v25n2.pdf
- See also: Validation of the automatic blood pressure monitor for children and adolescents — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0066-782X2009000100003
- See also: Validation of the Baecke questionaire for adolescents — http://www.scielo.mec.pt/pdf/rpcd/v6n3/v6n3a02.pdf
- Available data/document: Individual Participant Data Set — https://www.ncbi.nlm.nih.gov/pubmed/21874720 — The study by Bala and Drid (2010) was used for the sample calculation of the participants.